CLINICAL TRIAL: NCT03467009
Title: Bullying Prevention Intervention for Adolescent Primary Care Patients
Acronym: iPACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R21HD088739 (NIH); R21HD088739 (NIH)
Record Dates: First submitted 2018-02-27; First posted 2018-03-15 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-09

CONDITIONS: Cyberbullying
Keywords: cyber-victimization; text message; mhealth
MeSH Terms: conditions — Cyberbullying

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- iPACT Intervention (Experimental): 1. In-clinic brief session, introducing basic principles of cognitive behavioral theory and the structure of the text-message portion of the intervention.
  2. Eight-week longitudinal tailored CBT-based text-message program.
  Interventions: Behavioral: iPACT Intervention
- Control: Enhanced Usual Care (EUC) (Active Comparator): The investigators will provide participants with a standard resource sheet with information on bullying and mental health resources.
  Interventions: Other: Control: Enhanced Usual Care (EUC)
- iPACT Intervention- App (Experimental): 1. In-clinic brief session, introducing basic principles of cognitive behavioral theory and the structure of the message portion of the intervention delivered via app.
  2. Eight-week longitudinal tailored CBT-based message program delivered via app.
  Interventions: Behavioral: iPACT Intervention- app

INTERVENTIONS:
Behavioral: iPACT Intervention — Brief in-person + tailored, daily 8-week text-message secondary prevention intervention.
  Arms: iPACT Intervention
Other: Control: Enhanced Usual Care (EUC) — EUC group participants will receive standardized information on cyberbullying.
  Arms: Control: Enhanced Usual Care (EUC)
Behavioral: iPACT Intervention- app — Brief in-person + tailored, daily 8-week message secondary prevention intervention delivered via app.
  Arms: iPACT Intervention- App

SUMMARY:
The purpose of this randomized controlled study is to evaluate acceptability and feasibility, and to gather preliminary data about efficacy, of "iPACT" (intervention to Prevent Adolescent Cyber-victimization with Text messages), a brief in-clinic introductory session + longitudinal automated text-message-based secondary prevention program for adolescents with a history of past-year cyber-victimization presenting to a pediatric clinic for well-child visits.

DETAILED DESCRIPTION:
Cyber-victimization predicts depressive symptoms and suicidality; it correlates with PTSD symptoms, alcohol and other drug use, physical peer violence, and dating violence.

Almost 80% of adolescents have a well-child visit with their pediatrician each year. Pediatricians recognize this visit as an important opportunity for behavioral screening, interventions, and referrals, but they currently lack cyber-victimization interventions that are feasible and effective in the clinical setting. Personalized text-message interventions are accessible, feasible, and may be effective with these adolescents.

The purpose of this study is to test the feasibility and acceptability of a novel text-message-augmented secondary prevention intervention, "iPACT." Drawing on effective cognitive behavioral therapy (CBT) and motivational interviewing (MI) depression and violence prevention interventions, a brief in-clinic session will introduce basic cognitive and behavioral strategies. Following their clinic visit, eight weeks of tailored CBT-informed daily text messages will be sent, to enhance skills and remind participants of self-determined goals.

Participants will be identified in the course of usual clinical care. If eligible, parents will be consented and participants assented. Participants will complete a baseline assessment and will be randomized to experimental (iPACT, n=25) or enhanced usual care (EUC, n=25) care, using stratified block randomization.

iPACT group participants will participate in a brief, structured in-clinic introduction on CBT and the iPACT program, followed by 8 weeks of tailored, two-way, CBT-and MI-informed automated text messages (short message service, SMS). EUC group participants will receive standardized information on cyberbullying. The current standard of care for these patients is no care: no cyber-victimization screening assessment protocols are currently used in our clinic. Both iPACT and EUC conditions therefore exceed current levels of care.

At baseline, 8 week follow-up, and 16 week follow-up, participants will complete assessments on cyberbullying, peer violence, and cognitive/behavioral skill-sets. At the 8-week follow-up, standardized qualitative and quantitative process measures will be administered to assess efficacy, acceptability, usability, and feasibility.

ELIGIBILITY:
Inclusion Criteria:

* presenting to Hasbro Children's pediatric clinic
* being mentally and physically able to assent
* being English-speaking
* having a consentable parent present
* self-reporting cyber-victimization (defined as endorsing >1 past-year episode of technology-mediated victimization)

Exclusion Criteria:

* being cognitively or emotionally unable to take part in the intervention as determined by the pediatric attending clinician
* suspected by clinical staff of being a victim of child abuse
* currently incarcerated or under police custody

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 77 (Actual)
Dates: Start 2018-03-06 (Actual); Primary Completion 2019-06-12 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Intervention Acceptability: Enrollment Rate | Enrollment
  Enrollment Rate: % of eligible participants who consented and completed enrollment
Intervention Acceptability: Change in Follow Up Rate from 8 weeks post-enrollment to 16 weeks post-enrollment | 8 weeks post-enrollment (close of intervention), 16 weeks post-enrollment (8 wks after close of intervention)
  Retention Rate: % of consented participants who completed follow up
Intervention Acceptability: Participant Satisfaction | 8 weeks post-enrollment (close of intervention)
  Text Customer Satisfaction Questions
Intervention Feasibility: Participant Engagement | Enrollment to 8 weeks post-enrollment (close of intervention)
  Among the intervention group, how many participants responded to at least one of the daily text message queries, and how many requested on-demand support text-messages.

SECONDARY OUTCOMES:
Change in cyber-victimization between enrollment, 8 weeks post-enrollment, and 16 weeks post-enrollment | Enrollment, 8 weeks post-enrollment (close of intervention), 16 weeks post-enrollment
  Modified version of the University of New Hampshire Internet Safety Education Survey (Jones et al. 2012); investigators selected 5 items from the survey to measure. Items are scored by participants' self-report of online harassment experiences ranging from 0 ("Never") to 4 ("7 or more times"). Possible score range of 0-20, with higher scores indicating greater number of online harassment experiences.
Change in cyber-victimization emotional impact between enrollment, 8 weeks post-enrollment, and 16 weeks post-enrollment | Enrollment, 8 weeks post-enrollment (close of intervention), 16 weeks post-enrollment
  Modified version of the Cyber-Victimization Emotional Impact Scale (Elipe et al. 2015); investigators selected 7 of the 18 items to measure. Items are scored by participants' self-report of feelings ranging from 0 ("Not at all") to 4 ("Extremely"). Possible score range of 0-28, with higher scores indicating greater degree of emotional impact.
Change in cyber-victimization related behaviors between enrollment, 8 weeks post-enrollment, and 16 weeks post-enrollment | Enrollment, 8 weeks post-enrollment (close of intervention), 16 weeks post-enrollment
  Comprised of 5 items from the Bystander Intervention in Bullying Measures (Nickerson et al. 2014) and 8 items from the University of New Hampshire Internet Safety Education Survey (Jones et al. 2012). Items are scored by participants' self-report of online bystander behavior ranging from 1 ("Strongly disagree") to 5 ("Strongly agree"). Possible score range of 13-65, with higher scores indicating greater personal responsibility/self-efficacy to intervene when witnessing online harassment experiences.

CONTACTS AND LOCATIONS:
Overall Officials: Megan L Ranney, MD MPH, Principal Investigator — Rhode Island Hospital
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No